CLINICAL TRIAL: NCT03240523
Title: A Randomized, Parallel-group, Multicenter Study to Assess the Efficacy and Safety of Vilaprisan in Subjects With Uterine Fibroids
Brief Title: A Study to Assess Safety and Efficacy of Vilaprisan in Subjects With Uterine Fibroids
Acronym: ASTEROID 5
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Due to a change in the development program, the study was closed prematurely.
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15789; 2016-002855-48 (EudraCT Number)
Record Dates: First submitted 2017-07-21; First posted 2017-08-07 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Uterine Fibroids
MeSH Terms: conditions — Leiomyoma | interventions — vilaprisan

STUDY DESIGN:
Masking Description: With protocol version 5.0 the blinded study arms A3 and B were converted to one open-label study arm called A3/B.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A1: Vilaprisan (3/1 regimen) (Experimental): Orally, 2 mg, once daily, 3 months treatment followed by 1 menstrual bleeding episode
  Interventions: Drug: Vilaprisan (BAY1002670)
- Group A2: Vilaprisan (6/2 regimen) (Experimental): Orally, 2 mg, once daily, 6 months treatment followed by 2 menstrual bleeding episodes
  Interventions: Drug: Vilaprisan (BAY1002670)
- Group A3/B (3/2 regimen) (Experimental): Orally, 2 mg, once daily, 3 months treatment followed by 2 menstrual bleeding episodes
  With protocol version 5.0 the blinded study arms A3 and B were converted to one open-label study arm called A3/B.
  Interventions: Drug: Vilaprisan (BAY1002670)

INTERVENTIONS:
Drug: Vilaprisan (BAY1002670) — Orally, 2 mg, once daily

SUMMARY:
The primary objective of this study is to describe the efficacy of vilaprisan in subjects with uterine fibroids compared to ulipristal.

The secondary objective of this study is to evaluate the efficacy and safety of different treatment regimens of vilaprisan in subjects with uterine fibroids.

ELIGIBILITY:
Inclusion Criteria:

* Women, 18 years or older at the time of Visit 1
* Diagnosis of uterine fibroid(s) documented by ultrasound at screening with at least 1 fibroid with largest diameter more than 30 mm and less than 120 mm
* Heavy menstrual bleeding (HMB) >80.00 mL documented by menstrual pictogram (MP) in a bleeding episode period during the screening period
* Use of an acceptable non-hormonal method of contraception
* An endometrial biopsy performed during the screening period, without significant histological disorder such as endometrial hyperplasia (including simple hyperplasia) or other significant endometrial pathology

Exclusion Criteria:

* Pregnancy or lactation (less than 3 months since delivery, abortion, or lactation before start of treatment)
* Hypersensitivity to any ingredient of the study drugs
* Hemoglobin values ≤6 g/dL or any condition requiring immediate blood transfusion (subjects with hemoglobin values ≤10.9 g/dL will be recommended to use iron supplementation)
* Any diseases, conditions, or medications that can compromise the function of the body systems and could result in altered absorption, excessive accumulation, impaired metabolism, or altered excretion of the study drug including
* Abuse of alcohol, drugs, or medicines (eg: laxatives)
* Undiagnosed abnormal genital bleeding
* Any diseases or conditions that might interfere with the conduct of the study or the interpretation of the results

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 766 (Actual)
Dates: Start 2017-07-31 (Actual); Primary Completion 2020-06-28 (Actual); Study Completion 2021-10-25 (Actual)

PRIMARY OUTCOMES:
Amenorrhea (yes/no) | At 3 months (at the end of treatment perid 1)
  Defined as menstrual blood loss (MBL) < 2 mL based on the menstrual pictogram (MP) during last 28 days.
  For the primary analysis of the primary variable, the amenorrhea rates after 12 weeks of treatment in Groups A1, A2 and A3 will be compared to the rate from Group B.

SECONDARY OUTCOMES:
Total volume of menstrual blood loss | After approximately 1 year in subgroup 1 and after approximately 2 years in subgroup 2
  Assessed by menstrual pictogram (MP). Volume of menstrual blood loss will be normalized by 28 days.
Number of bleeding days | After approximately 1 year in subgroup 1 and after approximately 2 years in subgroup 2
  From day 1 of the first treatment period until the day before the next treatment period after the last treatment period would start again normalized to 28 days.
Amenorrhea (yes/no) | At 6 months, at 12 months, at 15 months, at 18 months, at 21 months and at 24 months
  Defined as menstrual blood loss (MBL) < 2 mL based on the menstrual pictogram (MP) during last 28 days of the treatment period.
Absence of bleeding (spotting allowed) | Up to 24 months
  Absence of bleeding defined as no bleeding (spotting allowed) during the last 28 days of the treatment; based on the UF-DBD (Uterine Fibroid Daily Symptom Diary).
Time to onset of controlled bleeding | Quarterly up to 24 months
  Onset of controlled bleeding is defined by the first day, for which the menstrual blood loss (assessed by MP) for all subsequent 28-day periods up to the end of the treatment period is less than 80.00 mL.
HMB (Heavy Menstrual Bleeding) responder rate | By treatment period up to 24 months
  Percentage of subjects with blood loss < 80.00 mL per 28 days and 50% reduction compared to baseline [assessed by MP]
Percent change in volume of largest fibroid compared to baseline | At baseline, at 12 months and at 24 months
  Measured by MRI (magnetic resonance imaging).
Endometrial histology | Up to 24 months
  E.g., benign endometrium, presence or absence of hyperplasia or malignancy
Endometrial thickness | Up to 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (139):
- Australia (4):
  - Paratus Clinical Pty Ltd, Blacktown, New South Wales
  - Paratus Clinical Wyong Complex, Kanwal, New South Wales
  - Women's Health and Research Institute of Australia-WHRIA, Sydney, New South Wales
  - Greenslopes Private Hospital, Greenslopes, Queensland
- Austria (3):
  - Medizinische Universität Graz, Graz, Styria
  - Landeskrankenhaus Bregenz, Bregenz, Vorarlberg
  - Universitätsklinikum AKH Wien, Vienna
- Belgium (6):
  - AZ Jan Palfijn Gent, Ghent, Oost-Vlaanderen
  - CHU Saint-Pierre/UMC Sint-Pieter, Bruxelles - Brussel
  - CU Saint-Luc/UZ St-Luc, Bruxelles - Brussel
  - CHU de Tivoli, La Louvière
  - CHR de la Citadelle - Department of Gynaecology & Obstetrics, Liège
  - Femicare vzw, Tienen
- Bulgaria (11):
  - MHAT Blagoevgrad AD, Blagoevgrad
  - MHAT Dobrich, Dobrich
  - MC Asklepii OOD, Dupnitsa
  - Multiprofile Hospital for Active Treatment Uni Hospital OOD, Panagyurishte
  - MHAT Avis Medika, Pleven
  - Spec. Hospital for Active Treatment of Oncological Diseases, Sofia
  - DCC Aleksandrovska, Sofia
  - Medical Center Panaceya, Sofia
  - MHAT Niamed, Stara Zagora
  - Multiprofile Hospital for Active Treatment Sv. Anna, Varna
  - SHOGAT Prof Dimitar Stamatov, Varna
- Canada (7):
  - Ocean West Research Clinic Inc, Surrey, British Columbia
  - Strand Clinic, St. John's, Newfoundland and Labrador
  - Ottawa Hospital-Riverside Campus, Ottawa, Ontario
  - Clinique OVO, Montreal, Quebec
  - Clinique Recherche en Sante des Femmes Inc., Québec
  - Centre de recherche Saint-Louis, Québec
  - ALPHA Recherche Clinique, Québec
- Czechia (8):
  - Fakultni nemocnice Brno, Brno
  - Gynekologicka ordinace - Ceske Budejovice, České Budějovice
  - G-Centrum Olomouc s.r.o. Dr. Skrivanek, Olomouc
  - MUDr. Martina Maresova Rosenbergova, gynekologie, Pilsen
  - Centrum gynekologicke rehabilitace, Písek
  - Dr. Smrhova-Kovacs, Tábor
  - MediGyn s.r.o., Třeboň
  - GYNEKO spol. s r.o., Vsetín
- Denmark (4):
  - Aarhus Universitetshospital, Skejby, Aarhus N
  - Nordsjælland Hospital Hillerød, Hillerød
  - Hvidovre Hospital, Hvidovre
  - Odense Universitetshospital, Gynækologisk Obstetrisk Afd. D, Odense C
- Finland (6):
  - HUS / Naistenklinikka, Helsinki
  - VL-Medi Oy, Helsinki
  - Kymenlaakson keskussairaala, Kotka
  - Lääkäriasema Cantti Oy, Kuopio
  - Lääkärikeskus Gyneko, Oulu
  - Turun yliopistollinen keskussairaala, Turku
- Germany (4):
  - Praxisklinik am Rosengarten, Mannheim, Baden-Wurttemberg
  - Frauenarztpraxis Dr. Wolfgang Clemens, Stolberg, North Rhine-Westphalia
  - Praxis f. Gynäkologie und Geburtshilfe, Bernburg, Saxony-Anhalt
  - emovis GmbH, Berlin
- Hungary (9):
  - Principal SMO Kft., Baja
  - Dr. Rethy Pal Korhaz - Rendelointezet Bekescsaba, Békéscsaba
  - Tritonlife Robert Magankorhaz, Budapest
  - Szent Anna szuleszeti-nogyogyaszati maganrendelo, Debrecen
  - NAP - Rendelo, Private Clinic, Debrecen
  - Debreceni Egyetem Klinikai Kozpont, Debrecen
  - Komaromi Selye Janos Korhaz, Komárom
  - SzSzBMK es EOK Josa Andras Oktatokorhaz, Nyíregyháza
  - SZTE ÁOK Szent Györgyi Albert Klinikai Kozpont, Szeged
- Midland Regional Hospital, Mullingar, Westmeath, Ireland
- Italy (4):
  - A.O.U. Policlinico G.Rodolico-San Marco, Catania, Sicily
  - A.O. Ospedali Riuniti Villa Sofia-Cervello, Palermo, Sicily
  - A.O.U. Careggi, Florence, Tuscany
  - A.O.U.I. Verona, Verona, Veneto
- Lithuania (6):
  - Jsc "Vakk", Kaunas
  - Klaipeda City Outpatient Clinic, Klaipėda
  - JSC Seimos gydytojas family medical center, Vilnius
  - JSC Gyvenk Silciau Medical Center Maxmeda, Vilnius
  - Private hospital and outpatient clinic "Kardiolita", Vilnius
  - Vilnius University Hospital Santaros Klinikos, Vilnius
- Netherlands (3):
  - Flevoziekenhuis, Almere Stad
  - VUmc, Amsterdam
  - Maasstad Ziekenhuis | Neurology Department, Rotterdam
- Norway (5):
  - Kirkeparken Spesialistpraksis, Fredrikstad
  - Nesttun Spesialistpraksis AS, Nesttun
  - Medicus Oslo AS, Oslo
  - Stavanger Universitetssjukehus, Stavanger
  - Medicus AS, Trondheim
- Poland (12):
  - Tomaszewski Medical Center, Bialystok
  - Prywatna Klinika Ginekologiczno-Poloznicza, Bialystok
  - CLINICAL MEDICAL RESEARCH Sp. z o. o., Katowice
  - Vita Longa Sp. z o.o., Katowice
  - Medico Praktyka Lekarska, Krakow
  - Prywatny Gabinet Lekarski Ginekologia, Poloznictwo i Ultr., Lodz
  - Centrum Medyczne Chodzki, Lublin
  - Specjalistyczny Gabinet Ginekologiczno-Polozniczy, Lublin
  - NZOZ NOVITA, Specjalistyczne Gabinety Lekarskie S.C, Lublin
  - VitroLive Sp. z o.o., Szczecin
  - NZOZ Zieniewicz Medical, Warsaw
  - Centrum Badawcze Wspolczesnej Terapii, Warsaw
- Portugal (3):
  - Centro Clinico Academico - Braga, Braga
  - CHUC - Hospitais da Universidade de Coimbra, Coimbra
  - Centro Hospitalar de Lisboa Ocidental | Clin Res Dept, Lisbon
- Slovakia (6):
  - Univerzitna nemocnica Bratislava, Nemocnica Ruzinov, Bratislava
  - ULMUS, s r.o., Hlohovec
  - GA Lucenec s.r.o, Lučenec
  - Galipea s.r.o., Nitra
  - Gyncentrum Nitra s.r.o., Nitra
  - Virina sano, s.r.o. Gynekologicko porodnicka ambulancia, Veľký Krtíš
- South Korea (13):
  - Dongguk University Ilsan Hospital, Goyang-si, Gyeonggido
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggido
  - Ajou University Hospital, Suwon, Gyeonggido
  - Inje University Haeundae Paik Hospital, Busan
  - Keimyung University Dongsan Medical Center, Daegu
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - Kangnam Sacred Heart Hospital, Seoul
  - CHA Gangnam Medical Center, Seoul
  - The Catholic University of Korea Seoul St. Mary's Hospital, Seoul
  - Korea University Guro Hospital, Seoul
  - Ewha Womans University Hospital, Seoul
- Spain (7):
  - Hospital Sanitas La Zarzuela, Aravaca, Madrid
  - Hospital de Basurto, Bilbao, Vizcaya
  - Hospital Universitario 12 de Octubre, Madrid
  - Ginemed, Seville
  - H Virgen del Rocio |Cardiology|AF|Stroke prevention, Seville
  - Hospital General Universitario de Valencia, Valencia
  - Hospital Universitario de Álava - Sede Txagorritxu, Vitoria-Gasteiz, Álava
- Sweden (4):
  - Södersjukhuset AB, Stockholm
  - Karolinska Universitetssjukhuset i Solna, Stockholm
  - Danderyds sjukhus, Stockholm
  - Akademiska Sjukhuset, Uppsala
- Taiwan (8):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - China Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Mackay Memorial Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Chang Gung Memorial Hospital at Linkou, Taoyuan District
- United Kingdom (5):
  - North Hampshire Hospital, Basingstoke, Hampshire
  - North Middlesex University Hospital, London
  - Whittington Hospital, London
  - Chelsea & Westminster Hospital, London
  - St Mary's Hospital (London), London

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.

REFERENCES:
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe — http://www.clinicaltrialsregister.eu/
- See also: Click here to find information for studies related to Bayer products. To find this study enter the ClinicalTrials.gov identifier (NCT) number or Bayer Study Identifier (ID) in the search field. — http://clinicaltrials.bayer.com